CLINICAL TRIAL: NCT02420405
Title: Mutation Detection of Small Specimens Obtained by Endobronchial Ultrasound Transbronchial Needle Aspiration in Advanced Nonsquamous Non-small Cell Lung Cancer Using Next-generation Sequencing
Brief Title: Mutation Detection of EBUS-TBNA Specimens Using NGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiayuan Sun (Other)
Responsible Party: Sponsor-Investigator, Jiayuan Sun, Director, Endoscope Department, Shanghai Chest Hospital, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHCHE201502
Record Dates: First submitted 2015-03-25; First posted 2015-04-17 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Lung Cancer
Keywords: Gene testing; Endobronchial ultrasound (EBUS); Next-generation sequencing (NGS); Small biopsies
MeSH Terms: conditions — Lung Neoplasms | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Routine gene testing (Placebo Comparator): Routine gene testing of EGFR, ROS1 and ALK will be performed on those diagnosed with nonsquamous NSCLC.
  Interventions: Procedure: Routine gene testing
- Next-generation sequencing (Experimental): Routine gene testing was performed in those diagnosed with nonsquamous NSCLC. NGS will be performed on these that have adequate rest tissues.
  Interventions: Procedure: Next-generation sequencing

INTERVENTIONS:
Procedure: Routine gene testing — For those diagnosed with nonsquamous NSCLC, routine gene testing including EGFR, ROS1 and ALK will be performed.
  Arms: Routine gene testing
Procedure: Next-generation sequencing — For those diagnosed with nonsquamous NSCLC and have done routine gene testing, NGS will be perform on those that have adequate rest tissues.
  Arms: Next-generation sequencing

SUMMARY:
The objective of the study was to compare the value of routine gene testing and next-generation sequencing (NGS) in detecting gene mutations of small specimens obtained by endobronchial ultrasound transbronchial needle aspiration (EBUS-TBNA) and get the knowledge of how many EBUS-TBNA samples were adequate for NGS.

DETAILED DESCRIPTION:
Some gene mutations can direct individualized treatment. The routine gene testing of EGFR, ROS1 and ALK is direct sequencing, Reverse transcription quantitative real-time polymerase chain reaction (RT-QPCR) and fluorescent in situ hybridization (FISH) or immunohistochemistry (IHC). Next-generation sequencing (NGS) is a new technique, which is more sensitive than routine techniques. So we decided to compare the value of gene testing between routine method and NGS in EBUS-TBNA specimens and get the knowledge of how many EBUS-TBNA samples were adequate for NGS.

The study was designed as a prospective and single center study. Seventy patients will be enrolled into the study and the clinical data of the patients, including his smoke history, cancer history, occupation exposure and so on, will be collected and recorded in a case report form. For the patients recruited in the study, the lymph nodes suspected to be malignant will be obtained by EBUS-TBNA. Samples will be sent to Pathology Department of Shanghai Chest Hospital and will be processed with paraffin-embedded, and for those diagnosed with nonsquamous NSCLC, routine gene testing of EGFR, ROS1 and ALK will be performed. And the rest tissues will be extracted with DNA and performed gene mutations using NGS for these qualified DNA samples.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are suspected with nonsquamous non-small cell lung cancer according to the clinical, lab examination and imaging data and had never been diagnosed as primary lung cancer before will be enrolled into the study.
2. The clinical stage of the patients should be in stage IIIA-IV judged by the imaging data and can't receive surgery initially.

4. There exist at least one lesions that can be obtained by EBUS-TBNA.

Exclusion Criteria:

1. The patient is highly suspected to benign lesion, small cell lung cancer and squamous cell carcinoma according to the clinical data.
2. Surgery was considered to be the primary treatment.
3. Patients who are diagnosed with lung cancer and received treatment with drugs or recurrent with lung cancer will be excluded.
4. Severe cardiopulmonary dysfunction and other indications that can't tolerate bronchoscopy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Values of gene testing between routine method and NGS in EBUS-TBNA specimens | Up to one and a half years

SECONDARY OUTCOMES:
The quantity of EBUS-TBNA samples adequate for NGS. | Up to one and a half years

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD,PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Heijden EH, Casal RF, Trisolini R, Steinfort DP, Hwangbo B, Nakajima T, Guldhammer-Skov B, Rossi G, Ferretti M, Herth FF, Yung R, Krasnik M; World Association for Bronchology and Interventional Pulmonology, Task Force on Specimen Guidelines. Guideline for the acquisition and preparation of conventional and endobronchial ultrasound-guided transbronchial needle aspiration specimens for the diagnosis and molecular testing of patients with known or suspected lung cancer. Respiration. 2014;88(6):500-17. doi: 10.1159/000368857. Epub 2014 Nov 5. PMID 25377908
- [Background] Wahidi MM, Herth F, Yasufuku K, Shepherd RW, Yarmus L, Chawla M, Lamb C, Casey KR, Patel S, Silvestri GA, Feller-Kopman DJ. Technical Aspects of Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration: CHEST Guideline and Expert Panel Report. Chest. 2016 Mar;149(3):816-35. doi: 10.1378/chest.15-1216. Epub 2016 Jan 12. PMID 26402427
- [Background] Folch E, Yamaguchi N, VanderLaan PA, Kocher ON, Boucher DH, Goldstein MA, Huberman MS, Kent MS, Gangadharan SP, Costa DB, Majid A. Adequacy of lymph node transbronchial needle aspirates using convex probe endobronchial ultrasound for multiple tumor genotyping techniques in non-small-cell lung cancer. J Thorac Oncol. 2013 Nov;8(11):1438-1444. doi: 10.1097/JTO.0b013e3182a471a9. PMID 24128714
- [Background] Coco S, Truini A, Vanni I, Dal Bello MG, Alama A, Rijavec E, Genova C, Barletta G, Sini C, Burrafato G, Biello F, Boccardo F, Grossi F. Next generation sequencing in non-small cell lung cancer: new avenues toward the personalized medicine. Curr Drug Targets. 2015;16(1):47-59. doi: 10.2174/1389450116666141210094640. PMID 25495923
- [Background] Marchetti A, Del Grammastro M, Filice G, Felicioni L, Rossi G, Graziano P, Sartori G, Leone A, Malatesta S, Iacono M, Guetti L, Viola P, Mucilli F, Cuccurullo F, Buttitta F. Complex mutations & subpopulations of deletions at exon 19 of EGFR in NSCLC revealed by next generation sequencing: potential clinical implications. PLoS One. 2012;7(7):e42164. doi: 10.1371/journal.pone.0042164. Epub 2012 Jul 27. PMID 22848739